CLINICAL TRIAL: NCT01462539
Title: Factors That Increase Length of Stay After Outpatient Surgery of 3-6 Year Olds With OSAS Symptoms Versus Without OSAS Symptoms After Adenotonsillectomy
Brief Title: Adenotonsillectomy and Obstructive Sleep Apnea Study
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB11-00364
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Adenotonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSAS group
- Non-OSAS group

SUMMARY:
Adenotonsillectomies are one of the most common childhood surgeries and are first-line treatment to correct childhood obstructive sleep apnea syndrome (OSAS). This is a study comparing patients with and without OSA looking at the length of stay following adenotonsillectomy and the factors affecting length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. history of snoring/gasping/ or pause in breathing reported by caregivers.
2. age 3-6 years old
3. undergoing adenotonsillectomy only no concurrent surgery
4. scheduled as outpatient and plan for discharge home

Exclusion Criteria:

1. Preoperatively requiring additional respiratory support
2. scheduled for concurrent surgery that could increase total general anesthetic time
3. recurrent adenotonsillitis as sole indication for surgery

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing adenotonsillectomy only with no concurrent surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS) | 1 Day (Day of Surgery)

SECONDARY OUTCOMES:
Cause of increased Length of stay (LOS) | 1 Day (Day of Surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Raman, MD, Principal Investigator — Nationwide Childrens Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States